CLINICAL TRIAL: NCT03773458
Title: Validation of the Utility of an Artificial System for the Large-scale Screening of Scoliosis Using Back Images
Brief Title: Validation of the Utility of an Artificial System for the Large-scale Screening of Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCPMOH2018-China-13
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Orthopedic Disorder of Spine; Artificial Intelligence; Scoliosis
Keywords: Orthopedic Disorder of Spine
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients for AI test. (Other): Device: An artificial system for the screening of scoliosis
  Interventions: Device: An artificial system for the screening of scoliosis

INTERVENTIONS:
Device: An artificial system for the screening of scoliosis — An artificial intelligence to make evaluation of scoliosis using back images

SUMMARY:
Traditional school scoliosis screening approaches remains debatable due to unnecessary referal and excessive cost. Deep learning algorithms have proven to be powerful tools for the detection of multiple diseases; however, the application of such methods in scoliosis screening requires further assessment and validation. Here, the investigators develop an artificial system for the automated screening of scoliosis using disrobed back images, and conduct clinical trial to validate if the diagnostic system can offsetting the shortcomings of human doctors.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients included both pretreatment back photos and whole spine (C7-S1) standing X-ray or ultrasound images (for healthy population); 2. All the documents are clear to be recognized by naked eyes; 3. Back photos and are taken at the same time (not >1month); 4.Patients were consider as idiopathic scoliosis according to clinical photos.

Exclusion Criteria:

* 1. Patients were considered as non-idiopathic scoliosis for obvious abnormal features of trunck,such as Cafe-au-Lait spots for neurofibromatosis, Spider finger, Abnormal hair spot of back, pelvic tilt, lower limb discrepancy and so on; 2.The taken time between back photo and X-ray or ultrasound was more than 1month; 3.The clinical photos and images were not clear; 4. The X-ray film or ultrasound images not including whole spine (C7-S1).

Ages: 10 Years to 22 Years | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
The proportion of accurate, mistaken and miss detection of the intelligent visual acuity diagnostic system. | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China